CLINICAL TRIAL: NCT03934515
Title: Tracheal etCO2 Level and Gastric pH Level Measurements During the Correct Naso-gastric Tube Placement in Unconscious Patients. A Physiological, Prospective, Observational Study
Brief Title: End-Tidal CO2 (etCO2) and pH in the Correct Naso-gastric Tube Placement
Acronym: NGT
Status: Completed | Type: Observational
Sponsor: Clinica Luganese Moncucco (Other)
Collaborators: Ospedale Regionale Bellinzona e Valli (Other)
Responsible Party: Principal Investigator, Samuele Ceruti, Principal Investigator, Clinica Luganese Moncucco
Other Study IDs: CLM_ICU_001
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Gastric Feeding Tube; Blood Gas Monitoring, Transcutaneous; pH
Keywords: naso-gastric tube, etCO2, pH
MeSH Terms: interventions — Hydrogen-Ion Concentration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - etCO2: At the end of the anaesthesia , as usual, the secretions are aspirated with a suction tube of 18 Fr of caliber (diameter 6 mm). When the tube is inserted into the endotracheal tube, before proceeding with the aspiration of the secretions, a capnometer is attached to its outer end, measuring the etCO2 value for 10-15 seconds. At the end of the measurement, authors proceed with the aspiration of the secretions as usual.
  Authors then proceed with the laying of a NGT according to local protocols. Also in this case, once the NGT has been inserted, the etCO2 is measured at the end of the probe for 10-15 seconds. At the end of the measurement, the capnometer can be detached, as a standard procedure, and the NGT can be used as usual.
  At the end of the procedure, therefore, for each patient, two values of etCO2 are acquired which will allow to obtain two "populations of values" of the etCO2: the values recorded at the endotracheal level and the one recorded at the oesophageal level.
  Interventions: Other: etCO2
- Group B - pH: At the end of the anaesthesia , once the NGT is inserted, the pH is measured by aspirating the gastric contents and measuring on specific litmus paper the pH values, both at a distance of 25 cm from the mouth (oesophageal site) and at a distance of 40 cm (gastric site).
  At the end of the procedure, for each patient two values of pH are acquired which will allow to obtain two pH "value populations": a value at oesophageal level and a value at the gastric level.
  Interventions: Other: pH

INTERVENTIONS:
Other: etCO2 — At the end of the procedure, therefore, for each patient two values of etCO2 are acquired which will allow to obtain two "populations of values" of the etCO2: the values at the endotracheal level and the esophageal level values. The authors will find the "threshold value" of etCO2 collected when the NGT is well positioned in trachea. The study manager is not directly involved in the measurement and recording of etCO2 values.
  Other Names: Group A
  Groups: Group A - etCO2
Other: pH — At the end of the procedure, for each patient two values of pH are acquired which will allow to obtain two pH "value populations": a value at esophageal level and a value at the gastric level. The authors will find the "threshold value" of pH collected when the NGT is positioned in the esophagus and in the stomach. The study manager is not directly involved in the measurement and recording of pH values.
  Other Names: Phase B
  Groups: Group B - pH

SUMMARY:
The laying of a naso-gastric tube is an extremely common event in intensive medicine; although standard naso-gastric tube laying is performed at the patient's bedside, this procedure is not without risk. Through the use of methods already used in the clinical field, of daily use, we want to identify the threshold value between tracheal and esophageal etCO2 (group A) and the threshold value between gastric and esophageal pH (group B).

DETAILED DESCRIPTION:
Numerous methodologies have been evaluated to recognize the correct positioning of NGT at the gastric level, including different clinical techniques (such as gastric auscultation, aspiration of the NGT), ultrasound techniques, etc. Actually, the diagnostic gold standard is the thoraco-abdominal anterior-posterior radiography, which is considered the only non-invasive method capable to confirm the correct pose of the NGT at intra-diaphragmatic level. This method, however, even if it is non-invasive, requires the use of ionizing radiation (4 micro-Sievert (uSv) for radiography) which could be repeated multiple time for the same patient; NGT may need to be repositioned several times during the same hospital stay, increasing patient exposure to ionizing radiation and, potentially, also the health workers exposure.

The aim is to identify into the group A the threshold value between tracheal and esophageal etCO2 and into the group B the theshold value between gastric and esophageal pH.

Phase A: etCO2 measurement will be collected 1. after intubation, when the tube is inserted into the endotracheal tube, before proceeding with the aspiration of secretions and 2. once the NGT has been inserted, by a probe located at the end of the tube.

Phase B: pH measurement will be collected at the end of the procedure, once the NGT is inserted, at 1.a distance of 25 cm from the mouth (oesophageal site) and at 2. a distance of 40 cm (gastric site), aspirating the gastric contents and measuring on specific litmus paper.

ELIGIBILITY:
Inclusion criteria:

* Adult patients (> 18 years)
* Patients male and female
* Patients intubated by oro- or naso-tracheal way
* Post-induction curarized patients
* Fasting patients (from at least 6 hours)

Exclusion criteria:

* Patient refusal
* Patients with known bleeding diathesis / ongoing bleeding
* Patients at risk of bleeding (defined as thrombocytes <50 G/l, fibrinogen <1.0 g/l, international normalized ratio (INR) > 2.5, activated partial thromboplastin time (aPTT) > 70 sec)
* Patients with traumatic brain injury / Polytrauma
* Patients with esophagus-tracheal fistulas or malformations of the ear, nose, and throat (ENT) sphere
* Patients with current or previous radiotherapy of the ENT sphere
* Patients unable to give their informed consent due to language barriers
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who required a NGT placement in Clinica Luganese Moncucco and in Regional Hospital of Bellinzona who will signed the Informed Consent Form
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
etCO2 level | 30-60 seconds
  to find a threshold value of etCO2 collected when the NGT is well positioned in trachea
pH | 30-60 seconds
  to find a threshold value of pH collected when the NGT is positioned in the esophagus and in the stomach.

SECONDARY OUTCOMES:
etCO2 level in chronic obstructive pulmonary disease (COPD) patients | 30-60 seconds
  subanalysis for the threshold value in the group with chronic obstructive pulmonary disease (COPD)
pH in patients taking proton pump inhibitors (PPIs) | 30-60 seconds
  identify patients taking proton pump inhibitors (PPIs) and perform a sub-subanalysis for the threshold value in the group with already diagnosed gastro-esophageal reflux disease.

CONTACTS AND LOCATIONS:
Overall Officials: Samuele Ceruti, MD, Principal Investigator — Clinica Luganese Moncucco
Locations (1):
- Clinica Luganese Moncucco, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bercik P, Schlageter V, Mauro M, Rawlinson J, Kucera P, Armstrong D. Noninvasive verification of nasogastric tube placement using a magnet-tracking system: a pilot study in healthy subjects. JPEN J Parenter Enteral Nutr. 2005 Jul-Aug;29(4):305-10. doi: 10.1177/0148607105029004305. PMID 15961688
- [Background] Nguyen L, Lewiss RE, Drew J, Saul T. A novel approach to confirming nasogastric tube placement in the ED. Am J Emerg Med. 2012 Oct;30(8):1662.e5-7. doi: 10.1016/j.ajem.2011.09.010. Epub 2011 Nov 17. PMID 22100480
- [Background] Ozer S, Benumof JL. Oro- and nasogastric tube passage in intubated patients: fiberoptic description of where they go at the laryngeal level and how to make them enter the esophagus. Anesthesiology. 1999 Jul;91(1):137-43. doi: 10.1097/00000542-199907000-00022. PMID 10422939
- [Background] Prasad G, Garg R. The 'bubble technique': an innovative technique for confirming correct nasogastric tube placement. J Clin Anesth. 2011 Feb;23(1):84-5. doi: 10.1016/j.jclinane.2010.03.006. No abstract available. PMID 21296259
- [Background] Vigneau C, Baudel JL, Guidet B, Offenstadt G, Maury E. Sonography as an alternative to radiography for nasogastric feeding tube location. Intensive Care Med. 2005 Nov;31(11):1570-2. doi: 10.1007/s00134-005-2791-1. Epub 2005 Sep 20. PMID 16172849
- [Result] Chun DH, Kim NY, Shin YS, Kim SH. A randomized, clinical trial of frozen versus standard nasogastric tube placement. World J Surg. 2009 Sep;33(9):1789-92. doi: 10.1007/s00268-009-0144-x. PMID 19626360
- [Result] Fernandez RS, Chau JP, Thompson DR, Griffiths R, Lo HS. Accuracy of biochemical markers for predicting nasogastric tube placement in adults--a systematic review of diagnostic studies. Int J Nurs Stud. 2010 Aug;47(8):1037-46. doi: 10.1016/j.ijnurstu.2010.03.015. PMID 20399427
- [Result] Gilbertson HR, Rogers EJ, Ukoumunne OC. Determination of a practical pH cutoff level for reliable confirmation of nasogastric tube placement. JPEN J Parenter Enteral Nutr. 2011 Jul;35(4):540-4. doi: 10.1177/0148607110383285. Epub 2011 May 27. PMID 21622643
- [Result] Kim HM, So BH, Jeong WJ, Choi SM, Park KN. The effectiveness of ultrasonography in verifying the placement of a nasogastric tube in patients with low consciousness at an emergency center. Scand J Trauma Resusc Emerg Med. 2012 Jun 12;20:38. doi: 10.1186/1757-7241-20-38. PMID 22691418
- [Derived] Ceruti S, Dell'Era S, Ruggiero F, Bona G, Glotta A, Biggiogero M, Tasciotti E, Kronenberg C, Lollo G, Saporito A. Nasogastric tube in mechanical ventilated patients: ETCO2 and pH measuring to confirm correct placement. A pilot study. PLoS One. 2022 Jun 2;17(6):e0269024. doi: 10.1371/journal.pone.0269024. eCollection 2022. PMID 35653380
- See also: Principles for medical research involving human subjects — https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- See also: Federal law concerning research on human subjects — https://www.admin.ch/opc/de/classified-compilation/20061313/index.html
- See also: Guideline for good clinical practice — https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e-6-r2-guideline-good-clinical-practice-step-5_en.pdf
- See also: Ordinance on Clinical Trials in Human Research — https://www.admin.ch/opc/de/classified-compilation/20121176/index.html